CLINICAL TRIAL: NCT02821104
Title: Complement and Cardiovascular Risk in Adolescents
Acronym: CCRIA
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Robert Hoffman, Professor, Ohio State University
Other Study IDs: Peds34
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Results first posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Cardiovascular Disease; Type 2 Diabetes
Keywords: Complement; endothelial function; insulin sensitivity; adolescents; inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2; Insulin Resistance; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Adolescents: Healthy non Hispanic white adolescents

SUMMARY:
This study evaluates how genetic variations in complement, a part of the immune system, affect cardiovascular risk in adolescents.

DETAILED DESCRIPTION:
Cardiometabolic diseases usually do not produce significant mortality and morbidity until adulthood. There is clear evidence, however, that these diseases have their origins in childhood and adolescence. With the rising incidence of obesity associated with poorer eating and less physical activity in children and adolescents it is important that the investigators study these diseases early in their course if the investigators are to prevent future cardiometabolic disease. While obesity clearly increases cardiometabolic risk, not all obese subjects are at increased risk; approximately 25-30% of obese adults and adolescents are metabolically healthy. The complement system is key physiological component in controlling inflammation and recent studies have indicated complement plays an important role in increasing obesity and cardiometabolic risk. Adults with proven cardiometabolic disease or at future risk for cardiometabolic disease have increased levels of the complement components C3, C3a-desArg, and C4 compared to healthy, not at risk, control subjects, independent of obesity. Increased C3 or C3a-desArg levels in adolescents are associated with increased cardiometabolic risk independent of obesity. Two specific single nucleotide polymorphisms (SNPs) in the intron for C3, rs11569562 and rs2250656, both with A>G polymorphisms, are associated with increased serum C3 levels, and increases in a variety of cardiovascular risk factors. No one has investigated how C3 polymorphisms affect risk factors in adolescents. The C4 gene has significant copy number variation and increased copy number is associated with increased C4 levels. The relationship of C4 gene copy number to cardiometabolic risk has not been studied in adults or adolescents. The short-term objectives of this study are to explore differences in cardiometabolic risk factors in overweight and obese adolescents with C3 polymorphisms and also to explore how C4 gene copy number variation affects risk factors. The investigators overall hypothesis is that variations in C3 polymorphisms, C4 gene copy number or both will have significant impact on cardiometabolic health in overweight and obese adolescents. Both traditional and nontraditional cardiometabolic risk markers, including measures of body habitus, blood pressure, lipids, vascular function, insulin secretion and sensitivity, inflammation, and clotting will be investigated in 100 overweight and obese adolescents. The investigators proposed study will help us understand the role of complement and its genetics in the development of cardiometabolic risk and in potentially developing genetic biomarkers for adolescents at increased risk.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adolescents age 12 to 18 years
* Medication free for 2 weeks except oral contraceptives in females
* Non Hispanic white

Exclusion Criteria:

* Chronic medications except for contraceptives in females.
* History of autoimmune disease either endocrine or connective tissue type
* History of hematologic or renal disease, malignancy or other chronic disease
* Hispanic ethnicity,
* African-American or Asian race

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy adolescents
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2016-06; Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Clinical Trials.gov

REFERENCES:
- [Derived] Hoffman RP, Copenhaver MM, Zhou D, Yu CY. Oral glucose tolerance response curve predicts disposition index but not other cardiometabolic risk factors in healthy adolescents. J Pediatr Endocrinol Metab. 2021 Apr 5;34(5):599-605. doi: 10.1515/jpem-2020-0619. Print 2021 May 26. PMID 33818037

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Adolescents: Healthy non-Hispanic white adolescents between 12 and 18 years of age
Period: Overall Study
Arm/Group | Healthy Adolescents
Started | 77
Completed | 77
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Non-Hispanic, healthy White adolescents
Groups:
- Healthy Adolescents: Healthy non-Hispanic white adolescents between 12 and 18 years
Arm/Group | Healthy Adolescents
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.2 (1.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 75
  More than one race | 0
  Unknown or Not Reported | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.0 (5.8)

OUTCOME MEASURES:

1. Primary Outcome: Complement C3 Genotype
Description: Genetic C3F genotype allele presence
Time Frame: Baseline
Population: Total population
Measure: Count of Participants; unit: Participants
Groups:
- Healthy Adolescents: Non Hispanic white
Arm/Group | Healthy Adolescents
Number analyzed (Participants) | 75
Participants
  FS | 22
  SS | 45
  FF | 2
  missing | 6

2. Primary Outcome: C4 Copy Number
Description: C4A or C4B gene copy numbers
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Adolescents
Number analyzed (Participants) | 75
Participants
  C4A Copy number: 1 | 14
  C4A Copy number: 2 | 35
  C4A Copy number: 3 | 15
  C4A Copy number: 4 | 6
  C4A Copy number: missing | 5
  C4A Copy number: 0 | 0
  C4B copy number: 1 | 20
  C4B copy number: 2 | 45
  C4B copy number: 3 | 3
  C4B copy number: 4 | 0
  C4B copy number: missing | 5
  C4B copy number: 0 | 2

3. Secondary Outcome: BMI
Description: Body mass index
Time Frame: Baseline
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | Healthy Adolescents
Number analyzed (Participants) | 75
kg/m^2 | 22.0 (0.7)

4. Secondary Outcome: Waist Circumference
Description: Waist circumference at narrowest point
Time Frame: Baseline
Measure: Mean (Standard Error); unit: cm
Arm/Group | Healthy Adolescents
Number analyzed (Participants) | 74
cm | 72.5 (1.5)

5. Secondary Outcome: Body Fat
Description: Percent body fat BodPod
Time Frame: Baseline
Measure: Mean (Standard Error); unit: percentage of total body weight
Arm/Group | Healthy Adolescents
Number analyzed (Participants) | 74
percentage of total body weight | 23.9 (1.2)

6. Secondary Outcome: Endothelial Function
Description: reactive hyperemia response to upper arm occlusion
Time Frame: 8 min
Measure: Mean (Standard Error); unit: percentage change from baseline FVR
Arm/Group | Healthy Adolescents
Number analyzed (Participants) | 72
percentage change from baseline FVR | -81.7 (0.9)

7. Secondary Outcome: Vascular Stiffness
Description: augmentation index of reflected blood pressure wave
Time Frame: baseline
Measure: Mean (Standard Error); unit: percentage of peak blood pressure
Arm/Group | Healthy Adolescents
Number analyzed (Participants) | 72
percentage of peak blood pressure | -3.3 (2.5)

8. Secondary Outcome: Endothelin 1
Time Frame: baseline
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Healthy Adolescents
Number analyzed (Participants) | 70
pg/ml | 2.06 (0.06)

9. Secondary Outcome: Inflammation
Description: IL6
Time Frame: baseline
Measure: Mean (Standard Error); unit: mg/ml
Arm/Group | Healthy Adolescents
Number analyzed (Participants) | 70
mg/ml | 0.68 (0.08)

10. Secondary Outcome: Clotting
Description: PAI1
Time Frame: baseline
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Healthy Adolescents
Number analyzed (Participants) | 70
pg/ml | 3.78 (0.32)

11. Secondary Outcome: Insulin Sensitivity
Description: Oral glucose tolerance test
Time Frame: baseline
Measure: Mean (Standard Error); unit: units
Arm/Group | Healthy Adolescents
Number analyzed (Participants) | 69
units | 4.25 (0.27)

ADVERSE EVENTS:
Time Frame: 4 hours
Arm/Group | Healthy Adolescents
All-Cause Mortality (participants affected / at risk) | 0/75
Serious Adverse Events (participants affected / at risk) | 0/75
Other Adverse Events (participants affected / at risk) | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT02821104/Prot_SAP_000.pdf
  • Informed Consent Form (2016-12-06): https://cdn.clinicaltrials.gov/large-docs/04/NCT02821104/ICF_001.pdf